CLINICAL TRIAL: NCT06174714
Title: Effectiveness of Indo-SURFT in Reducing Addictive Substance Use in Women With Substance Use Disorders: a Pilot Study
Brief Title: Effectiveness of Indo-SURFT in Reducing Addictive Substance Use in Women With Substance Use Disorders
Acronym: Indo-SURFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kristiana Siste, Dr. dr. Kristiana Siste, SpKJ(K) - Head of Department of Psychiatry, Faculty of Medicine, Indonesia University, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KET-735-2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MI and Indo-SURFT (Experimental): once a week motivational interviewing/motivational enhancement therapy (MI) for 4 weeks, followed by once a week CBT using Indonesia Substance Use Reduction for Female Therapy (Indo-SURFT) for 8 weeks.
  Interventions: Behavioral: Indonesia Substance Use Reduction for Female Therapy (Indo-SURFT)

INTERVENTIONS:
Behavioral: Indonesia Substance Use Reduction for Female Therapy (Indo-SURFT) — 4 weeks of motivational interviewing/motivational enhancement therapy (MI) followed by 8 weeks cognitive behavioral therapy (CBT) using Indo-SURFT module.

SUMMARY:
Relapse in women was associated with depression, interpersonal stress, and relationship conflict with others when compared with men. The differences in gender profiles with substance use disorders (SUD) leads to the need for management strategies that are sensitive to each gender. This is a challenge to build a new module that can be applied continuously by collaborating CBT and several other psychosocial interventions, such as motivational enhancement therapy. The investigators compiled Indonesia Substance Use Reduction for Female Therapy (Indo-SURFT). By implementing this module, it is hoped that it can provide short and long term effects and reduce the relapse rate in women with SUD.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-59 years old
* diagnosed with substance use disorders based on DSM-V or ICD-10

Exclusion Criteria:

* subjects with severe mental disorder or intellectual disability

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Abstinence from Substance Use | post-intervention (week 13)
  Timeline Follow Back (TLFB): to assess daily use of addictive substances by writing yes/no for 28 days. This data will be collected weekly retrospectively to reduce the risk of recall bias.
Decrease in Addiction Severity | pre-intervention (week 0), and post-intervention (week 13)
  Addiction Severity Index (ASI), Indonesia version, measuring several domains: 1) Medical health (n= 11), 2) Employment/ support status (n= 24), 3 & 4) Drug/ alcohol use (n= 35), 5) Illegal activity/ legal status (n= 32), 6) Family/ social relationships (n= 38) and 7) Psychiatric health (n= 23). Lesser score indicates better outcome.
Improvement in Motivation to Change | pre-intervention (week 0), and post-intervention (week 13)
  University of Rhode Island Change Assessment (URICA), measuring motivation to change with 4 domains: 1) pre-contemplation, 2) contemplation, 3) action, and 4) maintenance. A higher score indicates a better outcome.
Improvement in Substance Craving | pre-intervention (week 0), and post-intervention (week 13)
  Visual Analog Scale (VAS), measuring substance craving severity. Range 0 (no craving) - 100 (severe craving). A lower score indicates a better outcome.

SECONDARY OUTCOMES:
Improvement in Psychological Distress | pre-intervention (week 0), and post-intervention (week 13)
  Self-Report Questionnaire-20 (SRQ-20), measuring non-specific psychological distress. Score range 0-20; Scores >10 classified as mental distress. A lower score indicates a better outcome.
Improvement in Social Performance | pre-intervention (week 0), and post-intervention (week 13)
  Personal and Social Performance (PSP), measuring social function. A lower score indicates a better outcome.
Improvement in Quality of Life | pre-intervention (week 0), and post-intervention (week 13)
  World Health Organization Quality of Life (WHOQOL), measuring individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. A higher score indicates a better outcome.